CLINICAL TRIAL: NCT06315907
Title: Development and Validation of a Brief Food Noise Questionnaire
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, Corby K. Martin, Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2024-012
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Responses to survey questions — All 400 participants will first complete a demographic information survey and the new food noise questionnaire. Of these 400 participants, 250 participants will then complete additional questionnaires to assess construct validity. The remaining 150 participants will be asked to complete the food noise questionnaire again in approximately 1 week to assess test-retest reliability.

SUMMARY:
The purpose of the research is to develop and test the reliability and validity of a brief questionnaire to measure food noise.

DETAILED DESCRIPTION:
Currently and to our knowledge, there are no validated questionnaires to assess food noise. The purpose of this study is to develop and validate a brief food noise questionnaire. A total of 400 participants will be asked to complete the new food noise questionnaire. A subsample will also be asked to complete the questionnaire a second time to evaluate test-retest reliability. A separate subsample will also complete additional questionnaires to test convergent and discriminant validity.

ELIGIBILITY:
Inclusion Criteria:

* This study is open to adults (aged 18 years and above) who reside in the United States.

Exclusion Criteria:

* Individuals who do not provide informed consent will not progress to the survey questions
* Individuals who are currently participating in a weight loss program
* Individuals who have a BMI lower than 18.5 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be adults (18 years of age or older) residing in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants (N = 400) completed demographic information followed by the Food Noise Questionnaire (FNQ). This observational cohort study used a cross-sectional design to assess responses to the FNQ.
Period: Overall Study
Arm/Group | All Participants
Started | 400
Completed | 400
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 400 participants completed the online survey and demographic questions. Of these, 396 participants completed all Food Noise Questionnaire (FNQ) items and were included in the baseline analysis.
Arm/Group | All Participants
Number analyzed (Participants) | 396
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 309
  >=65 years | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266
  Male | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 48
  White | 286
  More than one race | 25
  Unknown or Not Reported | 26
Region of Enrollment [Number; unit: participants]
  United States | 396

OUTCOME MEASURES:

1. Primary Outcome: Scores on the Food Noise Questionnaire
Description: Food Noise Questionnaire (FNQ) measures persistent, intrusive thoughts about food that are disruptive to daily life and make healthy behaviors difficult. The FNQ consists of five items rated on a 5-point Likert scale: strongly disagree (scored as 0); disagree (scored as 1); neither agree nor disagree (scored as 2); agree (scored as 3); and strongly agree (scored as 4). A single total score for the questionnaire is calculated by summing responses for the five items. The total FNQ score ranges from 0 to 20, with higher total scores indicating greater levels of food noise.
Time Frame: The Food Noise Questionnaire (FNQ) was completed once as part of a larger online survey. The entire online survey was completed in approximately 30 to 45 minutes, and the FNQ items were completed in approximately 5 to 10 minutes.
Population: A total of 400 participants completed the online survey and demographic questions. Of these, 396 participants completed all Food Noise Questionnaire (FNQ) items and were included in the analysis of the outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 396
score on a scale | 7.39 (5.37)

ADVERSE EVENTS:
Time Frame: From the start to the end of the online survey session (approximately 30-45 minutes).
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/400
Serious Adverse Events (participants affected / at risk) | 0/400
Other Adverse Events (participants affected / at risk) | 0/400

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT06315907/Prot_SAP_000.pdf